CLINICAL TRIAL: NCT03170778
Title: Ocular and Vision Problems in Patients After Fontan Operation
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Susan Fernandes, Clinical Professor, Pediatrics - Cardiology Clinical Professor, Medicine - Cardiovascular Medicine, Stanford University
Other Study IDs: 36401
Record Dates: First submitted 2017-04-26; First posted 2017-05-31 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Congenital Heart Disease
Keywords: Congenital Heart Disease; CHD; Fontan
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purposes of this study are to identify indicators of vision problems and ocular abnormalities in patients with a Fontan circulation through a standardized questionnaire and to correlate the intraocular pressure measured with the Icare tonometer with central venous pressure measured with the VENUS 2000 CVP non-invasive system to determine whether intraocular pressure can be used as a surrogate measure of increased central venous pressure in patients with a Fontan circulation.

DETAILED DESCRIPTION:
Numerous authors have described optic disc edema, globe flattening, choroidal folds which were thought to be part of the well-defined but still idiopathic syndrome of idiopathic intracranial hypertension.

The pathogenesis of idiopathic intracranial hypertension is not well understood. Recent reports, however suggest that elevated cerebral venous pressure underlines the process. The close relationship that exist between spinal fluid pressure and cerebral venous pressure has been definitely established. It was found that patients with increased venous pressure due to heart failure had an increase in spinal fluid pressure as well.

Furthermore, numerous authors have described venous stasis retinopathy, bilateral choroidal detachments, intraretinal hemorrhages, vessel tortuosity, microaneurysms, capillary leakage, central retinal vein occlusion, open angle glaucoma, choroidal effusion, etc. in patients with pulmonary arterial hypertension. Elevated venous pressure found in pulmonary arterial hypertension is responsible for the delayed choroidal perfusion and the reduced venous blood outflow. This explains the clinical findings of venous stasis retinopathy, choroidal detachments, etc. which are related to elevated episcleral, retinal and choroidal venous pressure secondary to elevated systemic venous pressure (increased pulmonary vascular resistance in patients with pulmonary arterial hypertension leads to right heart failure and subsequent elevation in systemic venous pressure).

Systemic venous pressures in Fontan patients are comparable with those in patients with significant right heart failure in a 2- ventricular circulation. With Fontan anatomy the elevated central venous pressure is transmitted to the dural venous sinuses of the brain through jugular veins and the paraspinal venous plexus and after the Fontan procedure brain venous pressure are chronically elevated.

The investigators believe that the long-term effects of the Fontan operation can result in a spectrum of ocular changes similar to those occurring in patients with idiopathic intracranial and pulmonary arterial hypertensions due to chronically elevated cerebral venous pressure.

It has been reported that intraocular pressure is directly related to the episcleral and jugular venous pressure in patients without underlying ophthalmic diseases. Several previous studies have shown a linear correlation between central venous pressure and intraocular pressure. Therefore, the investigators believe that the monitoring of intraocular pressure may be simple and effective method for estimating central venous pressure in patients with Fontan circulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients (male and female) 18 and older with Fontan circulation

Exclusion Criteria:

* Patients under 18.
* Patients with any prior ocular trauma or surgery.
* Patients unwilling to consent to study.
* Patients who are unable to speak and read English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted solely in the the Adult Congenital Heart Clinic at Stanford, and patients with congenital heart disease (CHD) will be recruited for the study.
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2016-02-13 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Reported ocular medical history in Fontans | The final 3 months will be used for data analysis and the presentation/manuscript preparation.
  Number of participants with Fontan physiology that have undergone a Fontan operation that have reported any changes in ocular and vision abnormalities by using a standardized survey.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Fernandes, LPD, PA-C, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital Adult Congenital Heart Clinic, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No